CLINICAL TRIAL: NCT00000562
Title: Extracorporeal Support for Respiratory Insufficiency (ECMO)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 200; R01HL016154-05 (Other Grant/Funding Number: US NIH Grant Number)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2000-01

CONDITIONS: Acute Respiratory Failure; Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Extracorporeal Membrane Oxygenation

INTERVENTIONS:
Procedure: extracorporeal membrane oxygenation

SUMMARY:
To evaluate indications for the use and efficacy of extracorporeal membrane oxygenators (ECMO's) for the support of patients with potentially reversible acute respiratory failure.

DETAILED DESCRIPTION:
BACKGROUND:

The report of the Task Force on Respiratory Diseases identified a clinical syndrome of acute respiratory insufficiency (ARI) and estimated that approximately 60,000 Americans die of ARI yearly. ARI was not precisely defined; indeed, the Task Force realized that pathologists do not recognize ARI. The Task Force pointed out that no diagnostic tests for early detection of ARI exist, that the incidence and prevalence of the disease are not known, and that existing therapy is supportive and nonspecific (diuretics, corticosteroids, etc.). The pathogenesis of the syndrome, the mechanism of interstitial edema, the defenses of the lung against agents causing ARI, and the ultrastructural pathology and natural history of the disease were virtually unknown. The Task Force indicated a need for Respiratory Care Centers with highly trained personnel that could reduce mortality from ARI.

This clinical trial grew out of the Task Force report. Nine participating centers defined ARI in clinical and physiological terms and agreed to a prospective randomized study for 3 years to compare treatment of severe ARI by conventional means with treatment by extracorporeal membrane oxygenators.

Animal studies have shown that ECMO's can provide one to two weeks' support for the lungs without serious blood damage, in contrast to bubble oxygenators, which allow complete pulmonary bypass for approximately 6 hours, after which severe blood damage occurs at the direct blood-gas interface. If patients with hypoxia secondary to acute reversible lung injury can be supported with ECMO's until the lung lesion heals, improvement in survival rates and avoidance of the hazards of conventional therapy may result. The trial, now completed, was conducted at nine clinical centers in the United States.

DESIGN NARRATIVE:

Randomized, non-blind, fixed sample; 90 eligible patients were randomly assigned to a group receiving extracorporeal membrane oxygenation plus conventional therapy or to a group receiving conventional therapy.

The study completion date listed in this record was obtained from the Query/View/Report (QVR) System.

ELIGIBILITY:
Men and women, ages 12 to 65, not stratified as to ethnic group, who had potentially reversible acute respiratory failure.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1974-06; Study Completion 1979-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bartlett — University of California, Irvine; Philip Drinker — Brigham and Women's Hospital; L. Edmunds — University of Pennsylvania; Alan Morris — University of Utah; E. Pierce — Icahn School of Medicine at Mount Sinai; Herbert Proctor — University of North Carolina; Arthur Thomas — University of California; Warren Zapol — Massachusetts General Hospital

REFERENCES:
- [Background] National Heart, Lung, and Blood Institute, Extracorporeal Support for Respiratory Insufficiency, A Collaborative Study. December 1979.
- [Background] Zapol WM, Snider MT, Hill JD, Fallat RJ, Bartlett RH, Edmunds LH, Morris AH, Peirce EC 2nd, Thomas AN, Proctor HJ, Drinker PA, Pratt PC, Bagniewski A, Miller RG Jr. Extracorporeal membrane oxygenation in severe acute respiratory failure. A randomized prospective study. JAMA. 1979 Nov 16;242(20):2193-6. doi: 10.1001/jama.242.20.2193. PMID 490805